CLINICAL TRIAL: NCT05483127
Title: Clinical Comparison of Two Daily Disposable Toric Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLA306-P002
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Astigmatism; Ametropia; Myopia
Keywords: Contact lenses; Vision; Eye sight
MeSH Terms: conditions — Astigmatism; Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- P1fA, then MDT (Other): Verofilcon A toric soft contact lenses worn first, followed by stenfilcon A toric soft contact lenses, as randomized. Each study lens type will be worn for 8 (-0/+3) days for at least 10 hours per day. Lenses will be removed nightly and disposed of after a single use.
  Interventions: Device: Verofilcon A toric soft contact lenses; Device: Stenfilcon A toric soft contact lenses
- MDT, then P1fA (Other): Stenfilcon A toric soft contact lenses worn first, followed by verofilcon A toric soft contact lenses, as randomized. Each study lens type will be worn for 8 (-0/+3) days for at least 10 hours per day. Lenses will be removed nightly and disposed of after a single use.
  Interventions: Device: Verofilcon A toric soft contact lenses; Device: Stenfilcon A toric soft contact lenses

INTERVENTIONS:
Device: Verofilcon A toric soft contact lenses — Soft contact lenses for optical correction of ametropia and astigmatism
  Other Names: PRECISION1™ for Astigmatism; P1fA
Device: Stenfilcon A toric soft contact lenses — Soft contact lenses for optical correction of ametropia and astigmatism
  Other Names: MyDay® toric soft contact lenses; MDT

SUMMARY:
The primary purpose of this study is to demonstrate noninferiority in the visual acuity at distance when wearing PRECISION1™ for Astigmatism (P1fA) soft contact lenses compared to another commercially available, soft toric contact lens, MyDay® toric (MDT).

DETAILED DESCRIPTION:
Study participants will wear each study lens type in 1 of 2 randomized, crossover sequences. Participants will be expected to attend 4 visits and wear study lenses for at least 10 hours per day. The total duration of an individual's participation in the study will be up to 28 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wearers of toric soft contact lenses in both eyes with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.
* Able to wear contact lenses within a range of sphere & cylinder power and axes.
* Willing to NOT use rewetting/lubricating drops at any time during the study.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Current or previous P1fA and MDT habitual lens wearers.
* Monovision and multifocal lens wearers.
* Participation of the subject in a clinical trial within the previous 30 days or currently enrolled in any clinical trial.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (11):
- United States (11):
  - Kurata Eyecare Center, Los Angeles, California
  - Sabal Eye Care, Longwood, Florida
  - Drs. Giedd, P.A., Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Franklin Park Eye Center, Franklin Park, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - Heart of America Eye Care, P.A., Shawnee Mission, Kansas
  - Wesley Optometric Consulting, Medina, Minnesota
  - ProCare Vision Center, Granville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 11 investigative sites located in the United States.
Pre-assignment Details: Of the 153 enrolled, 1 participant was exited prior to randomization as a screen failure. This reporting group includes all randomized participants (152).
Groups:
- P1fA, Then MDT: Verofilcon A toric soft contact lenses worn first, followed by stenfilcon A toric soft contact lenses, as randomized. Each study lens type was worn for 8 (-0/+3) days for at least 10 hours per day. Lenses were removed nightly and disposed of after a single use.
- MDT, Then P1fA: Stenfilcon A toric soft contact lenses worn first, followed by verofilcon A toric soft contact lenses, as randomized. Each study lens type was worn for 8 (-0/+3) days for at least 10 hours per day. Lenses were removed nightly and disposed of after a single use.
Period: First Wear Period, 8 (-0/+3) Days
Arm/Group | P1fA, Then MDT | MDT, Then P1fA
Started | 77 | 75
Completed | 77 | 75
Not Completed | 0 | 0
Period: Second Wear Period, 8 (-0/+3) Days
Arm/Group | P1fA, Then MDT | MDT, Then P1fA
Started (One participant discontinued between First Wear Period and Second Wear Period due to an adverse event.) | 76 | 75
Completed | 76 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized subjects who are exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | P1fA, Then MDT | MDT, Then P1fA | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (9.4) | 34.3 (8.6) | 34.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 29 | 29 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 65 | 66 | 131
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 66 | 132
  Black or African American | 5 | 5 | 10
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 0 | 1
  Multi-Racial | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 77 | 75 | 152

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Means Distance Visual Acuity With Study Lenses at Week 1
Description: Distance visual acuity (VA) was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). A logMAR acuity of 0.0 corresponds to 20/20 Snellen (normal distance visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 8 of each study lens type worn during the corresponding crossover period
Population: Full Analysis Set with data at visit.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- PRECISION1 for Astigmatism (P1fA): Verofilcon A toric soft contact lenses worn during Period 1 or Period 2, as randomized. The study lenses were worn for 8 (-0/+3) days for at least 10 hours per day. Lenses were removed nightly and disposed of after a single use.
- MyDay Toric (MDT): Stenfilcon A toric soft contact lenses worn during Period 1 or Period 2, as randomized. The study lenses were worn for 8 (-0/+3) days for at least 10 hours per day. Lenses were removed nightly and disposed of after a single use.
Arm/Group | PRECISION1 for Astigmatism (P1fA) | MyDay Toric (MDT)
Number analyzed (Participants) | 151 | 151
Number analyzed (eyes) | 302 | 302
logMAR | -0.11 (0.005) | -0.10 (0.005)
Statistical Analysis 1: Comparison: PRECISION1 for Astigmatism (P1fA) vs MyDay Toric (MDT); Test type: Non-Inferiority — Noninferiority in distance VA was declared if upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least squares mean difference = -0.01, 95% CI 1-sided [upper limit -0.00], Standard Error of Mean 0.003 — LSM results based on mixed effects repeated measures model with both fixed (lens, visit, lens by visit interaction, period, sequence) and random (subject) effects. Difference=P1fA - MDT. Sign (negative or positive) is retained with the rounded value

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit, up to 28 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- P1fA Ocular; P1fA Non-Ocular: Events reported in this group occurred while exposed to the verofilcon A contact lenses.
- MDT Ocular; MDT Non-Ocular: Events reported in this group occurred while exposed to the stenfilcon A contact lenses.
Arm/Group | Pretreatment | P1fA Ocular | P1fA Non-Ocular | MDT Ocular | MDT Non-Ocular
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/304 | 0/152 | 0/302 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/304 | 0/152 | 0/302 | 0/151
Other Adverse Events (participants affected / at risk) | 0/152 | 0/304 | 0/152 | 0/302 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT05483127/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT05483127/SAP_001.pdf